CLINICAL TRIAL: NCT04616430
Title: Karma CREME-1: A Double-blind, Placebo-controlled, Three-armed, Pilot Study of the Effects, Safety and Tolerability of Topical Endoxifen in Women Within the Karma Cohort
Brief Title: Topical Endoxifen in Women
Acronym: CREME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Atossa Therapeutics, Inc. (Industry)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ATOS-010
Record Dates: First submitted 2020-10-16; First posted 2020-11-05 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Mammographic Breast Density
MeSH Terms: interventions — 4-hydroxy-N-desmethyltamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Topical Placebo:Transcutol™ (2-(2-Ethoxyethoxy)ethanol); isopropanol, Crodamol™ GTCC (a fully saturated emollient triester) and mineral oil
  Interventions: Drug: Placebo
- Topical Endoxifen 10mg/breast/day (Active Comparator): 10 mg/day topical (Z)-endoxifen; Transcutol™ (2-(2-Ethoxyethoxy)ethanol); isopropanol, Crodamol™ GTCC (a fully saturated emollient triester) and mineral oil
  Interventions: Drug: Topical endoxifen
- Topical Endoxifen 20mg/breast/day (Active Comparator): 20 mg/day topical (Z)-endoxifen; Transcutol™ (2-(2-Ethoxyethoxy)ethanol); isopropanol, Crodamol™ GTCC (a fully saturated emollient triester) and mineral oil
  Interventions: Drug: Topical endoxifen

INTERVENTIONS:
Drug: Topical endoxifen — topical solution
  Arms: Topical Endoxifen 10mg/breast/day; Topical Endoxifen 20mg/breast/day
Drug: Placebo — topical
  Arms: Control

SUMMARY:
Karma CREME-1 consisted of 90 participants from the Karma Cohort. The major focus of the pilot trial was to estimate time to mammographic density change. The primary objective was to determine the effect size of the breast density change between topical placebo and two doses of topical endoxifen.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the Karma Cohort
* Attending the national mammography screening program, i.e., aged 40-74 and have performed a screening mammogram maximum 3 months prior to study inclusion
* Mammographic density ~4.5 % density (volumetric) measured by Volpara, at the screening mammogram performed in connection to baseline (maximum 3 months prior to inclusion). The threshold value of 4.5% corresponds to the clinical Bl-RADS score A
* Postmenopausal, defined as no period of menstruation during last 12 months independent of any hormonal treatment
* Informed consent must be signed before any study specific assessments are performed

Exclusion Criteria:

* Any previous or current diagnosis of breast cancer (including carcinoma in situ).
* Any previous diagnosis of cancer with the exception of non-melanoma skin cancer and in situ cancer of the cervix.
* A history of major surgery of the breast, e.g., reduction or enlargement, which might affect density measurements.
* Mammographic Bl-RADS malignancy code 3, or above, at baseline mammography, or at mammography during time of treatment. Recall for additional examinations due to technical problems with the mammogram is accepted.
* Currently using estrogen and progesterone based hormone replacement therapy (oral or patches). Local estrogen treatment is accepted (ex. Vagifem).
* Non-medical approved drugs against hot-flashes including phytoestrogen.

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — heatlhy post-menopausal women
Enrollment: 90 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Hall, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sodersjukhuset, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Backlund M, Eriksson M, Gabrielson M, Hammarstrom M, Quay S, Bergqvist J, Hellgren R, Czene K, Hall P. Topical Endoxifen for Mammographic Density Reduction-A Randomized Controlled Trial. Oncologist. 2022 Jul 5;27(7):e597-e600. doi: 10.1093/oncolo/oyac102. PMID 35604960

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Topical Endoxifen 10mg/Breast/Day | Topical Endoxifen 20mg/Breast/Day
Started | 30 | 30 | 30
Completed | 23 | 2 | 0
Not Completed | 7 | 28 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Topical Endoxifen 10mg/Breast/Day | Topical Endoxifen 20mg/Breast/Day | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (6.01) | 56.9 (7.97) | 57.7 (8.41) | 56.5 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 30 | 90
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 30 | 30 | 30 | 90
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.9 (2.77) | 25.6 (3.57) | 25.2 (3.08) | 25.2 (3.1)
Blood pressure (systolic) [Mean (Standard Deviation); unit: mm Hg] | 117.5 (12.1) | 123.7 (8.45) | 120.4 (10.1) | 120.5 (10.5)
Weight [Mean (Standard Deviation); unit: kg] | 69.0 (7.33) | 69.8 (9.74) | 70.2 (9.31) | 69.7 (8.8)
Height [Mean (Standard Deviation); unit: cm] | 166.6 (5.14) | 165.3 (6.38) | 167.0 (6.06) | 166.3 (5.9)
Mammographic Breast Density [Mean (Standard Deviation); unit: % Dense Tissue] | 23.6 (17.2) | 23.9 (12.9) | 26.2 (18) | 24.6 (16.0)
Blood pressure (diastolic) [Mean (Standard Deviation); unit: mm Hg] | 77.0 (7.13) | 79.7 (5.86) | 77.0 (7.13) | 77.4 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mammographic Breast Density At Study Exit
Description: Change, on an individual level, in mammographic breast density, measured at 6 months or when exiting from the study (baseline screening mammography)
Time Frame: From baseline to study exit up to 6 months
Population: Due to dropouts, analysis could only be performed 1 time at study exit. Participants were encouraged to have a mammogram at study exit; not all did.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Control | Topical Endoxifen 10mg/Breast/Day | Topical Endoxifen 20mg/Breast/Day
Number analyzed (Participants) | 26 | 21 | 27
percent change from baseline | -1.85 (5.58) | -2.14 (6.50) | -3.75 (7.81)

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Control | Topical Endoxifen 10mg/Breast/Day | Topical Endoxifen 20mg/Breast/Day
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 27/30 | 28/30 | 27/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=30) | Topical Endoxifen 10mg/Breast/Day (N=30) | Topical Endoxifen 20mg/Breast/Day (N=30)
Rapid heart rate or palpitations (Cardiac disorders) | 13 (25) | 3 (4) | 4 (5)
Feel lightheaded (dizzy) (Ear and labyrinth disorders) | 14 (20) | 10 (15) | 4 (5)
Eyesight changes (Eye disorders) | 9 (15) | 5 (8) | 5 (7)
Constipation (Gastrointestinal disorders) | 3 (4) | 5 (7) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 3 (3) | 2 (2)
Difficulty swallowing (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 5 (6) | 3 (3) | 1 (2)
Feel bloated (Gastrointestinal disorders) | 13 (24) | 10 (13) | 4 (5)
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Burning feeling from breast tissue or breast skin (General disorders) | 6 (11) | 5 (8) | 7 (8)
Fragile mucous membranes (General disorders) | 18 (39) | 14 (22) | 14 (14)
Irritation from the breast skin (General disorders) | 8 (13) | 12 (14) | 15 (17)
Itching from the breast skin (General disorders) | 6 (14) | 21 (36) | 22 (36)
Lack of energy (General disorders) | 3 (6) | 6 (6) | 3 (3)
Pain (General disorders) | 4 (5) | 3 (3) | 1 (1)
Pain from breast tissue or breast skin (General disorders) | 3 (4) | 4 (7) | 3 (3)
Redness on breast skin (General disorders) | 4 (7) | 9 (10) | 9 (9)
Swelling of arms or legs (General disorders) | 2 (3) | 0 (0) | 0 (0)
Deviating lab value (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight gain (Investigations) | 15 (31) | 9 (14) | 4 (4)
Lack of appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Muscle cramps (e.g. in legs) (Musculoskeletal and connective tissue disorders) | 18 (38) | 11 (14) | 11 (14)
Pain in joints (Musculoskeletal and connective tissue disorders) | 14 (34) | 10 (16) | 11 (12)
Difficulty concentrating (Nervous system disorders) | 4 (4) | 0 (0) | 2 (2)
Feeling drowsy (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Headaches (Nervous system disorders) | 17 (31) | 11 (16) | 5 (6)
Numbness/tingling in the hands and feet (Nervous system disorders) | 5 (5) | 2 (2) | 2 (2)
Difficulty sleeping (Psychiatric disorders) | 13 (20) | 9 (9) | 4 (4)
Feeling nervous (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Feeling sad (Psychiatric disorders) | 4 (6) | 3 (4) | 2 (2)
Irritable (Psychiatric disorders) | 9 (22) | 10 (12) | 5 (6)
Mood swings (Psychiatric disorders) | 8 (21) | 9 (9) | 6 (6)
Sexual feeling decreased (Psychiatric disorders) | 23 (50) | 19 (28) | 15 (15)
Worry (Psychiatric disorders) | 6 (8) | 1 (1) | 0 (0)
Problems with urination (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Breast sensitivity/tenderness (Reproductive system and breast disorders) | 8 (13) | 8 (10) | 8 (8)
Dryness vaginal (Reproductive system and breast disorders) | 22 (46) | 22 (33) | 13 (14)
Menopausal hot flushes (Reproductive system and breast disorders) | 19 (48) | 14 (22) | 16 (17)
Night sweats (Reproductive system and breast disorders) | 21 (47) | 13 (19) | 14 (15)
Painful intercourse (Reproductive system and breast disorders) | 19 (41) | 16 (24) | 14 (15)
Vaginal bleeding or spotting (Reproductive system and breast disorders) | 1 (3) | 2 (2) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 10 (25) | 9 (12) | 4 (5)
Vaginal itching/irritation (Reproductive system and breast disorders) | 5 (12) | 6 (10) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 3 (5)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 5 (11) | 4 (6) | 3 (4)
Hair loss (Skin and subcutaneous tissue disorders) | 9 (19) | 9 (14) | 8 (8)
Itching (Skin and subcutaneous tissue disorders) | 4 (5) | 8 (10) | 12 (14)
Rashes on breast skin (Skin and subcutaneous tissue disorders) | 12 (24) | 21 (35) | 26 (43)
Skin rashes (Skin and subcutaneous tissue disorders) | 13 (20) | 13 (19) | 17 (22)

LIMITATIONS AND CAVEATS:
Early discontinuation of subjects due to AEs related to skin reactions lead to small numbers of completed subjects and inability to analyze the primary endpoint as outlined in the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT04616430/Prot_SAP_000.pdf